CLINICAL TRIAL: NCT04139993
Title: A Pilot Trial of Preoperative Oral Microbiota-Based Investigational New Drug, RBX7455 to Target Immune Response in Patients With Operable Stage I-III Breast Cancer
Brief Title: RBX7455 Before Surgery for the Treatment of Operable Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: poor accrual
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-004024; NCI-2021-02748 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19-004024 (Other: Mayo Clinic in Florida)
Record Dates: First submitted 2019-10-22; First posted 2019-10-25 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Breast Adenocarcinoma; Invasive Breast Carcinoma; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (RBX7455) (Experimental): Prior to standard of care surgery, patients receive RBX7455 orally (PO) 4 days a week for 2-4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Microbiota-based Formulation RBX7455

INTERVENTIONS:
Drug: Microbiota-based Formulation RBX7455 — Given PO
  Other Names: RBX 7455; RBX-7455; RBX7455

SUMMARY:
This clinical trial studies the side effects and possible benefits of RBX7455 given before surgery in treating patients with breast cancer that can be removed by surgery (operable). RBX7455 contains live intestinal microbes (active drug), which are obtained from healthy human stool and may restore the normal balance of microorganisms in the intestines through the transplant of live and beneficial microorganisms.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of microbiota-based formulation RBX7455 (RBX7455) given for at least 2 weeks and not more than 4 weeks prior to surgery.

II. To evaluate intratumoral immunomodulatory effects, including tumor infiltrating lymphocytes ( TILs), CD4, and CD8 T cells, in operable breast cancer patients.

SECONDARY OBJECTIVES:

I. To evaluate systemic immunomodulatory effects of RBX7455 by measuring circulating cytokines including IL-1b, IL-2, IL-4, IL-5, IL-6, IL-7, CXCL8 (IL-8), IL-10, IL-12, IL-13, IL- 17A, IFN-gamma, TNF-alpha, CCL2 (MCP-1), CCL4 (MIP-1beta), granulocyte-colony stimulating factor (G-CSF), and granulocyte macrophage (GM)-CSF before and after treatment with RBX7455.

II. To assess stool microbiome α-diversity, bacterial abundance, and bacterial taxonomy before and after treatment with RBX7455.

III. To assess the durability of bacterial engraftment of RBX7455 in the stool at 8 weeks and 6 months.

OUTLINE:

Prior to standard of care surgery, patients receive RBX7455 orally (PO) 4 days a week for 2-4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of surgery, patients are followed up at 8 weeks and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Histologically confirmed un-resected operable invasive adenocarcinoma of the breast >= 0.5cm

  * For cohort 1: Estrogen receptor (ER) and/or progesterone receptor (PR) positive >= 10%, and no human epidermal growth factor receptor 2 (HER2) amplification or overexpression
  * For cohort 2: Human epidermal growth factor receptor 2 (HER2) amplification with fluorescence in situ hybridization (FISH) ratio >= 2.0 or overexpression by immunohistochemistry 3+ with any ER and/or PR
  * For cohort 3: Triple negative. Estrogen receptor (ER) and/or progesterone receptor (PR) negative < 10%, and no human epidermal growth factor receptor 2 (HER2) amplification or overexpression
* Patients must not receive neoadjuvant chemotherapy prior to surgery
* Absolute neutrophil count (ANC) >= 1000/mm^3
* Platelet count >= 75,000/mm^3
* Hemoglobin >= 9.0 g/dL
* Creatinine =< 2 x upper limit of normal (ULN)
* Serum glutamic-oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 2 x ULN
* Albumin >= 3 g/dL
* Willing and able to swallow capsules
* Willing and able to complete the stool and serum testing required for the study
* Willing to provide blood samples for correlative research purposes
* Agrees not to take non-dietary probiotics through 8 weeks after receiving the course of study drug (including over-the counter [OTC] and prescription)
* Agrees not to take any oral vancomycin, metronidazole, fidaxomicin, rifaximin, nitazoxanide, bezlotoxumab and intravenous immunoglobulin therapy (IVIG) through the 8-week follow-up assessment unless newly prescribed by a treating investigator during the course of the study
* Willing to employ adequate contraception from the time of enrollment through 3 months after the final dose of RBX7455

  * Note: Adequate contraception methods include birth control pills, barrier device, intrauterine device
* Capable of understanding the investigative nature, potential risks, and benefits of the study
* Capable of providing valid informed consent
* Willing to return to enrolling institution for all study visits (blood draws, etc)
* Willing and able to complete the required Patient Medication Diary
* Willing and able to meet all study requirements, including attending all assessment visits and telephone calls
* Women of child bearing potential must have negative pregnancy test within 7 days of enrollment

Exclusion Criteria:

* Requires systemic antibiotic therapy for other condition
* Fecal microbiota transplant (FMT) within the past 6 months
* FMT with an associated serious adverse event related to the FMT product or procedure
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimen
* Immunocompromised patients including patients known to be human immunodeficiency virus (HIV) positive or those on chronic steroids > 20 mg prednisone a day or prednisone-equivalent

  * Note: Must be off systemic steroids at least 90 days prior to enrollment. However, topical steroids, inhalants or steroid eye drops are permitted
* Receiving any other investigational agent
* History of inflammatory bowel disease (IBD), e.g., ulcerative colitis, Crohn's disease, or microscopic colitis
* Diagnosis of irritable bowel syndrome (IBS) as determined by Rome III criteria
* History of chronic diarrhea
* History of celiac disease
* Currently has a colostomy
* Intraabdominal surgery related to gastrointestinal tract within the last 60 days
* Evidence of active, severe colitis
* History of short gut syndrome or motility disorders
* Requires the regular use of medications to manage bowel hypermotility
* Active autoimmune disease that has required systemic treatment in the =< 30 days (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs) prior to randomization. Note: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment. Patients with vitiligo, Graves' disease, or psoriasis not requiring systemic treatment within the past 30 days are not excluded
* Pregnancy
* Breast feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-01-11 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 4 weeks prior to surgery
  Assessed per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The maximum grade for each type of toxicity will be recorded for each patient, and frequency (percentage) of toxicity for all patients will be reported by study statistician and reviewed by primary disease site to determine toxicity patterns. Evaluation of RBX7455 will be assessed by physical exams and laboratory testing with number of patients with abnormal laboratory values and adverse events.

SECONDARY OUTCOMES:
Systemic immunomodulatory effects | Up t0 6 months after treatment
  The percent change in plasma concentrations of interleukin (IL)-1beta, IL-2, IL-4, IL-5, IL-6, IL-7, CXCL8 (IL-8), IL-10, IL-12, IL-13, IL-17A, IFN-gamma, TNF-alpha, CCL2 (MCP-1), CCL4 (MIP-1beta), granulocyte-colony stimulating factor (G-CSF), and granulocyte macrophage (GM)-CSF. will be summarized as mean (standard deviation) or median (range) where appropriate. Each of these factors will be plotted against time with the points belonging to a particular individual connected. Each graph will be visually inspected for trends across time and difference between treatment regimens. For each marker, the number of patients with at least a 2-fold increase/decrease in the number of cells/plasma concentration (marker specific response) after the first cycle of treatment as well as anytime during treatment will be determined.
Engraftment rate | Up to 6 months after treatment
Durability of bacterial engraftment of RBX7455 | Up to 6 months after treatment
  Will be evaluated with bacterial taxonomy using provided stool samples obtained by patient.

CONTACTS AND LOCATIONS:
Overall Officials: Maria I Vazquez Roque, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States